CLINICAL TRIAL: NCT01930968
Title: Use of Definity® Contrast Agent for Ultrasound of Intraocular Tumors
Brief Title: Definity for Ultrasound of Intraocular Tumors
Status: Withdrawn | Type: Observational
Why Stopped: Study did not receive funding to move forward
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Hans Grossniklaus, MD, Professor, Emory University
Other Study IDs: IRB00039493
Record Dates: First submitted 2013-02-28; First posted 2013-08-29 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Ocular Melanoma
Keywords: Uveal melanoma, ocular melanoma
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultrasound measurement: There is only 1 arm in this study. The ocular tumors will be imaged using ultrasound and the contrast agent. The patient's history will be noted, lung and heart auscultation will be performed, and blood pressure readings will be obtained to ensure the patient has no contraindications to using Definity®. If there are no contraindications, routine ocular ultrasonography, both A and B scans, will be performed using an Ellex Eye Cubed ultrasound machine. Definity® (the microbubble contrast agent) will be prepared per package instruction and the dose calculated according to the following formula: Patient weight (kg) X 10 microliters = Definity® dose. If necessary, a second 10 microliter/kg dose may be given 30 minutes after the first IV injection.

SUMMARY:
The study will test the usefulness of a contrast agent to help image tumors in the eye. In this study, patients with eye melanoma who are going to have their eye removed, will have their eye imaged by ultrasound (sound waves) before and after intravenous injection of microbubbles. The pathology characteristics of the tumor in the removed eye will be compared with the images.

DETAILED DESCRIPTION:
The investigators plan to enroll and image 10 patients with intraocular tumors who are going to undergo enucleation of their eye for the tumor. Definity®, a perflutren containing microsphere manufactured by Lantheus Medical Imaging, Inc., is commercially available and FDA approved for cardiac imaging. It is contraindicated for use in patients with pulmonary hypertension, unstable cardiopulmonary conditions, and cardiac shunts (right-to-left, bi-directional, or transient right-to left). After informed consent is obtained, a cardiologist will examine the patient's history, perform lung and heart auscultation, and obtain a blood pressure in order to ensure the patient has no contraindications to using Definity®. If there are no contraindications, routine ocular ultrasonography, both A and B scans, will be performed using an Ellex Eye Cubed ultrasound machine. Definity® will be prepared per package instructions and the appropriate dose will be calculated. If necessary, a second 10 microliter/kg dose may be give 30 minutes after the first IV injection. A bubble test (intravenous small amount of Definity injected with cardiac echo) will be performed in the cardiology imaging suite, clinical building A, in order to ensure that the patient does not have a right to left shunt. After that, Definity® will be administered as a slow IV bolus followed by a normal saline 10cc flush. The ultrasonographer will continue the ocular B scan during administration of Definity®. Vital signs will be obtained and documented at 30 minutes after administration of the last dose of Definity® and longer if needed.

ELIGIBILITY:
Inclusion Criteria:

* Adults 20 years old or over 18 years old with large uveal melanoma who are going to undergo enucleation

Exclusion Criteria:

* Patient with right-to-left, bi-direction, or transient right-to-left cardiac shunts
* Worsening of or clinically unstable congestive heart failure
* Acute myocardial infarctions or acute coronary syndromes
* Serious ventricular arrhythmias or high risk for arrhythmias, due to prolongation of the QT-interval (>60 msec)
* Respiratory failures marked by signs and symptoms of CO2 retention or hypoxemia
* Severe emphysema, pulmonary emboli, or other conditions that cause pulmonary hypertension due to compromised pulmonary-arterial vasculature
* Known hypersensitivity to perflutren (if the patient has been exposed to perflutren in the past and had an allergic reaction)
* Pregnancy or nursing mothers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over 20 years old with intraocular tumors (melanoma, metastasis, retinal tumors) who are going to undergo enucleation diagnosed in the Emory Eye Center Ocular Oncology Service. Patients will be assessed by a cardiologist or cardiology fellows.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Quantification of tumor perfusion and visualization of microvasculature using ultrasound enhanced images of intraocular tumors with microbubbles | Up to 2 years
  Ultrasound will be used to acoustically identify microbubbles in vascular channels in the intraocular tumors, including uveal melanoma, metastases and retinal tumors. Blood vessels in the tumor and retina are identified after IV injection of Definity® microbubbles which is used as the ultrasound contrast agent.

SECONDARY OUTCOMES:
Correlation between tumor vascularity by contrast enhanced ultrasoungraphy and histologically determined tumor vascular density | Up to 2 years
  The uptake of the Definity® microbubbles by the blood vessels in the tumor as determined by contrast enhanced ultrasoungraphy will be correlated with histologically determined tumor size and mean vascular density.
Correlation between tumor size by contrast enhanced ultrasoungraphy and histologically determined tumor size | Up to 2 years
  The tumor size as determined by contrast enhanced ultrasoungraphy will be correlated with histologically determined tumor size.

CONTACTS AND LOCATIONS:
Locations (1):
- Emory Eye Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Once research is completed, results of the study will be published in a specialty journal